CLINICAL TRIAL: NCT07289568
Title: Surgical Outcomes in Splenic Flexure Cancers: A Prospective, Multicentric Observational Cohort Study Comparing Segmental Hemicolectomy and Extended Hemicolectomy - The SPARROW Study
Brief Title: Surgical Outcomes in Splenic Flexure Cancers: A Multicenter Comparison of Segmental vs. Extended Hemicolectomy (SPARROW Study)
Acronym: SPARROW
Status: Enrolling by invitation | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025.249.IRB2.115
Record Dates: First submitted 2025-11-18; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Colon Cancer; Splenic Flexure Mobilization; Right Hemicolectomy; Left Hemicolectomy; Segmental Colectomy; Extended Hemicolectomy
Keywords: Splenic Flexure Cancer; Colorectal Cancer; Colon Adenocarcinoma; Overall Survival; Anastomotic Leak; Ileus; Postoperative Complications; Surgical Outcomes; Right Hemicolectomy; Left Hemicolectomy; Segmental Colectomy; Extended Hemicolectomy
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Anastomotic Leak; Ileus; Postoperative Complications | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colectomy — Extended hemicolectomy involves removal of a larger segment of colon that includes the splenic flexure tumor and its associated lymphatic drainage. The procedure typically includes ligation of the relevant feeding arteries-such as the right, middle, and left colic branches-and resection of adjacent colon segments to achieve an oncologically adequate specimen with tension-free anastomosis. The extent of resection and vascular ligation is determined according to surgeon preference and tumor location. This approach may be performed using open, laparoscopic, or robotic techniques, depending on institutional practice.
  Other Names: Extended Hemicolectomy; Segmental Colectomy

SUMMARY:
SPARROW Study: Surgical Outcomes in Splenic Flexure Cancer

Colonic cancers located at the splenic flexure where the transverse colon turns into the descending colon are uncommon and represent less than 10% of all colorectal cancers. Because of their unique location between the blood supply of the right and left colon, there is no clear agreement on which surgical method provides the best results.

Two main procedures are used:

Segmental hemicolectomy, which removes only the part of the colon containing the tumor, and

Extended hemicolectomy, which removes a larger section of the colon and more lymph nodes.

The SPARROW Study is a prospective, multicenter observational study designed to compare these two surgical approaches in patients with splenic flexure cancer. The study will include about 140 patients (70 in each group) from multiple tertiary colorectal centers in Turkey and Europe.

Researchers will collect information about each patient's surgery, recovery, and follow-up outcomes. The main outcomes include postoperative ileus, leakage at the surgical connection (anastomosis), wound infection, and total postoperative complications. Other outcomes include number of lymph nodes removed, complete tumor resection (R0), hospital stay, recovery time, reoperation, and 3-year overall and disease-free survival.

By analyzing both short- and long-term results, the SPARROW Study aims to provide high-quality evidence to guide surgeons in choosing the best and safest operation for patients with splenic flexure cancers.

All participants will provide written informed consent before joining the study. The study has received ethical approval from the Koç University Ethics Committee and will be conducted in accordance with the Declaration of Helsinki.

DETAILED DESCRIPTION:
Study Rationale:

Splenic flexure cancers pose unique surgical challenges due to their variable blood supply and lymphatic drainage. The optimal extent of resection remains controversial, with both extended right and left colectomy approaches showing different technical advantages. However, there are no prospective multicenter data comparing their perioperative and oncologic outcomes.

Study Design:

This is a prospective, multicenter observational cohort study involving tertiary colorectal cancer centers. The study will enroll 140 consecutive adult patients (≥18 years old) undergoing elective curative resection for histologically confirmed splenic flexure adenocarcinoma. Surgical approach-segmental or extended colectomy-will be chosen according to the operating surgeon's routine practice and preference, not assigned by randomization.

Primary Outcomes:

Postoperative ileus (incidence and duration)

Anastomotic leakage

Wound infection

Total postoperative complications

Secondary Outcomes:

Lymph node yield and R0 resection rate

Postoperative mortality

Operation time and estimated blood loss

Hospital stay, return to regular diet, and time to first flatus

Reoperation rates

3-year overall survival (OS) and disease-free survival (DFS)

Timeline:

Study start: 2025

Enrollment period: 24 months

Follow-up: 36 months per patient

Total duration: approximately 5 years

Ethical Conduct:

Ethical approval was obtained from the Koç University Ethics Committee. Each participating center will obtain local ethics approval. The study adheres to the principles of the Declaration of Helsinki and Good Clinical Practice (GCP).

Expected Impact:

This will be the first prospective multicenter observational study to compare segmental and extended hemicolectomy for splenic flexure cancers. The results will help standardize surgical decision-making and improve patient outcomes for this uncommon and technically challenging tumor location.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Histologically confirmed adenocarcinoma of the splenic flexure
* Elective surgical resection performed with curative intent (segmental colectomy or extended hemicolectomy)
* Availability of complete perioperative and follow-up data
* Written informed consent provided prior to participation
* Surgery performed by colorectal or general surgeons meeting institutional eligibility criteria (≥20 colorectal cancer cases/year, ≥2 years of colorectal training)

Exclusion Criteria:

* Emergency surgery for obstruction, perforation, or bleeding
* Non-adenocarcinoma histology (e.g., lymphoma, neuroendocrine tumor, gastrointestinal stromal tumor)
* Patients undergoing palliative resections, local excisions, or bypass procedures without curative intent
* Presence of synchronous colorectal malignancy or distant metastasis requiring simultaneous resection
* Previous colorectal resection involving the splenic flexure
* Patients with incomplete clinical or pathological data or those lost to follow-up before 30 days postoperatively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients diagnosed with splenic flexure adenocarcinoma who undergo elective curative resection (segmental or extended hemicolectomy) at participating tertiary colorectal surgery centers in Turkey and Europe. All patients will be treated according to the surgeon's standard practice and institutional protocols. Data will be collected prospectively for both perioperative and follow-up outcomes as part of the multicenter SPARROW Study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Ileus After Surgery for Splenic Flexure Cancer | Within 30 days after surgery
  The presence of postoperative ileus will be evaluated as the main indicator of early perioperative recovery. Ileus is defined as intolerance to oral intake and absence of bowel function beyond the expected postoperative period, requiring nasogastric decompression or delayed diet advancement. Data will be collected from medical records and postoperative progress notes. Additional related variables-such as the duration of ileus, need for nasogastric tube reinsertion, and time to first flatus-will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bilgi Baca, MD, Professor of Surgery, Principal Investigator — Acibadem University Istanbul Turkey
Locations (1):
- Acibadem University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be shared, including baseline demographic information, surgical approach (segmental vs. extended hemicolectomy), operative characteristics, short-term perioperative outcomes, and follow-up survival data. No directly identifiable information (such as names, contact details, or institutional identifiers) will be included. Data will be available in a secure, de-identified format for qualified researchers upon reasonable request to the SPARROW Study Steering Committee through the Turkish Society of Colon and Rectal Surgery (TKRCD), following approval of a data-use agreement and ethical review.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting materials will be available beginning 12 months after publication of the primary manuscript and will remain available indefinitely for qualified researchers upon reasonable request.
Access Criteria: Qualified researchers affiliated with academic institutions, professional societies, or healthcare organizations may request access to the de-identified dataset, study protocol, statistical analysis plan, and informed consent form. Requests should be submitted in writing to the SPARROW Study Steering Committee via the Turkish Society of Colon and Rectal Surgery (TKRCD). Access will be granted after approval of the research proposal and signing of a data-use agreement ensuring ethical conduct, confidentiality, and non-commercial use. Data will be shared electronically through a secure, password-protected institutional platform.

REFERENCES:
- [Result] Kuzu MA, Benlice C, Parvaiz A, Gorgun E, Bertelsen CA, Wexner S, Dozois EJ, Hohenberger W, Miskovic D, Sugihara K, Spinelli A, Wiggers T, Lee WY, Moslein G, Tsarkov P, Basany EE, Patron Uriburu JC, Perez RO, Lynch C, Liu Z, Hahnloser D, Nilsson PJ, Chowdri NA, Brown G, Rouanet P, Madoff RD, West NP, Sahin T, Elhan AH, Bordeianou LG; Colon Cancer Delphi Consensus Study Group. Standardizing the Definition of Each Colon Cancer Segment: Delphi Consensus on Clinical Decision-Making for Oncologic Outcomes. Dis Colon Rectum. 2025 Jul 1;68(7):835-844. doi: 10.1097/DCR.0000000000003739. Epub 2025 Apr 11. PMID 40214091
- [Result] Gebauer S, Schootman M, Xian H, Xaverius P. Neighborhood built and social environment and meeting physical activity recommendations among mid to older adults with joint pain. Prev Med Rep. 2020 Feb 11;18:101063. doi: 10.1016/j.pmedr.2020.101063. eCollection 2020 Jun. PMID 32140385
- [Result] Wang C, Wang C, Qiu J, Gao J, Liu H, Zhang Y, Han L. Ultrasensitive, high-throughput, and rapid simultaneous detection of SARS-CoV-2 antigens and IgG/IgM antibodies within 10 min through an immunoassay biochip. Mikrochim Acta. 2021 Jul 20;188(8):262. doi: 10.1007/s00604-021-04896-w. PMID 34282508
- [Result] Hohenberger W, Weber K, Matzel K, Papadopoulos T, Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation--technical notes and outcome. Colorectal Dis. 2009 May;11(4):354-64; discussion 364-5. doi: 10.1111/j.1463-1318.2008.01735.x. Epub 2009 Nov 5. PMID 19016817

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07289568/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT07289568/ICF_001.pdf